CLINICAL TRIAL: NCT02293863
Title: A Study of MHAA4549A in Combination With Oseltamivir Versus Oseltamivir in Participants With Severe Influenza A Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GV29216; 2014-000461-43 (EudraCT Number)
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Results first posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — gedivumab; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A: MHAA4549A 3600 mg + Oseltamivir (Experimental): Participants will receive a single low IV dose of MHAA4549A on Day 1 and standard oseltamivir therapy for minimum of 5 days.
  Interventions: Drug: MHAA4549A; Drug: Oseltamivir
- B: MHAA4549A 8400 mg + Oseltamivir (Experimental): Participants will receive a single high IV dose of MHAA4549A on Day 1 and standard oseltamivir therapy for minimum of 5 days.
  Interventions: Drug: MHAA4549A; Drug: Oseltamivir
- C: Placebo + Oseltamivir (Placebo Comparator): Participants will receive a single IV dose of placebo matched to MHAA4549A on Day 1 and standard oseltamivir therapy (75 or 150 mg BID) for minimum of 5 days.
  Interventions: Drug: Oseltamivir; Drug: Placebo

INTERVENTIONS:
Drug: MHAA4549A — Participants will receive a single dose of MHAA4549A by IV infusion on Day 1
  Arms: A: MHAA4549A 3600 mg + Oseltamivir; B: MHAA4549A 8400 mg + Oseltamivir
Drug: Oseltamivir — Participants will receive oseltamivir capsule either 75 mg or 150 mg BID orally for minimum of 5 days. Dosage and administration should follow local prescribing information for oseltamivir.
  Other Names: Tamiflu
Drug: Placebo — Participants will receive a single IV dose of placebo matched to MHAA4549A on Day 1
  Arms: C: Placebo + Oseltamivir

SUMMARY:
This is a randomized, double-blind, placebo-controlled study that will investigate the safety and clinical activity of a single intravenous (IV) dose of MHAA4549A in adult participants hospitalized with severe influenza A in combination with oseltamivir versus a comparator arm of placebo with oseltamivir.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of influenza A where a Sponsor-approved influenza test is used as an aid in diagnosis. A Sponsor-approved influenza test includes: Influenza antigen test or Influenza polymerase chain reaction (PCR) test
* One of the following markers of severity within 24 hours of admission: requirement for O2 supplementation to maintain SpO2 greater than (>) 92 %; or requirement for Positive Pressure Ventilation (PPV)
* A negative urine or serum pregnancy test for women of childbearing potential within 2 days prior to study treatment
* Participants of reproductive potential must agree to use acceptable contraceptive measures as per the protocol as a minimum, and local guidelines, if more stringent

Exclusion Criteria:

* Pregnant or lactating women, or women who intend to become pregnant during the study
* Hypersensitivity to monoclonal antibodies or any constituents (sodium succinate, sucrose, polysorbate 20) of study drug
* Hypersensitivity to the active substance or to any excipients of oseltamivir
* Investigational therapy within the 30 days prior to study treatment
* Received prior therapy with any anti-influenza monoclonal antibody therapy (including MHAA4549A) within 8 months prior to study treatment
* Current treatment (within 7 days of dosing) with probenecid, amantadine or rimantidine
* Participants who have taken more than a total of 6 doses (3 doses for peramivir) of anti-influenza therapy (e.g., oseltamivir, zanamivir, laninamivir, peramivir) in the period from onset of symptoms and prior to study treatment
* Admission >48 hours prior to study treatment
* Onset of influenza symptoms (including fever, chills, malaise, dry cough, loss of appetite, myalgias, coryza, or nausea) >5 days prior to study treatment
* Positive influenza B or influenza A + B infection within 2 weeks prior to study treatment
* High probability of mortality in the next 48 hours as determined by the investigator
* Participants requiring home or baseline oxygenation therapy
* Participants with history of chronic lung disease with a documented SpO2 less than (<) 95% off oxygen
* Participants on chronic dose of corticosteroids exceeding 10 milligrams per day (mg/day) of prednisone or equivalent steroid dose for duration of greater than 14 days within 30 days of entry into study
* Participants with the following significant immune suppression: bone marrow or solid organ transplant in the previous 12 months; cancer chemotherapy in the previous 12 months, HIV infection with most recent Cluster of Differentiation 4 (CD4) <200 cells per milliliter (cells/mL), or other significant immune suppression as determined by the investigator in discussion with the Sponsor Medical Monitor
* Participants on extracorporeal membrane oxygenation (ECMO) at time of randomization
* Any disease or condition that would, in the opinion of the site investigator or Sponsor, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (171):
- Belgium (4):
  - CHU St Pierre (St Pierre), Brussels
  - Hospital Erasme; Neurologie, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - CHU UCL Mont-Godinne, Mont-godinne
- Brazil (6):
  - Santa Casa de Misericordia; de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - PUC Campinas, Campinas, São Paulo
  - FUNFARME, São José do Rio Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz; Oncologia, São Paulo, São Paulo
  - Hospital Edmundo Vasconcelos, Vila Clementino, São Paulo
- Bulgaria (11):
  - MHAT "Dr. Tota Venkova"- Gabrovo, Gabrovo
  - University Multiprofile Hospital for Active Treatment "St. George", Plovdiv
  - SHATPPD Dr. Dimitar Gramatikov, Ruse Ltd., Rousse
  - Multiprofile Hospital for Active Treatment AKTA-MEDIKA EOOD, Sevlievo
  - MHAT Lyulin EAD, Department of internal diseases, Sofia
  - MHAT TOKUDA SOFIA/ICU-Intensive Care Unit, Sofia
  - 5th Multifunctional Hospital for Active treatment, Sofia
  - Military Medical Academy- MHAT, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov EAD, Sofia
  - MBAL St Marina Dep Pulmonology, ICU, Varna
  - Multiprofile District Hospital for Active Treatment Dr. Stefan Cherkezov AD, Veliko Tarnovo
- Canada (19):
  - Peter Lougheed Centre, Calgary, Alberta
  - Alberta Health Services, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia
  - Victoria General Hospital, Victora, British Columbia
  - Royal Jubilee Hospital Victoria general Hospital, Victoria, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - LHSC - University Hospital; Research Pharmacy, London, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Toronto East General, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre Hospitalier de la Universite Laval, Québec, Quebec
  - Pavillion Chul-Chuq, Sainte-Foy, Quebec
  - Centre de santé et de services sociaux de Trois-Rivières, Trois-Rivières, Quebec
- Chile (2):
  - Hospital Dr. Hernan Henriquez Aravena, Temuco
  - Clinica Renaca, Viña del Mar
- Czechia (5):
  - The University Hospital Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Anesthesia and Intensive Care Dept., Regional Hospital Liberec, Liberec
  - University hospital Ostrava, Clinic of infectious medicine, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Klinika anesteziologie a resuscitace, Prague
- France (13):
  - CH Victor Dupouy, Argenteuil
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - Service de Réanimation médicale - Bocage Central, Dijon
  - APHP Raymond Poincare, Garches
  - CHD Vendée, La Roche-sur-Yon
  - CHRU Lille, Lille
  - Réanimation Polyvalente, CHU Limoges, Limoges
  - CHRU Nancy, Nancy
  - Archet 1 university Hospital, Nice
  - HOPITAL COCHIN university hospital, Paris
  - Réanimation médicale NHC, Strasbourg
  - Hopital Universitaire Hautepierre, Strasbourg
  - Service de réanimation médicale, Hôpital Bretonneau, Tours
- Germany (5):
  - Uniklinik Köln, Medizinischen Klinik I, Cologne
  - Universitätsklinikum Frankfurt Goethe Universität, Frankfurt
  - Universitätsklinikum Heidelberg, Heidelberg
  - Uniklinikum Mainz, Mainz
  - Uniklinik Tübingen, Tübingen
- University of Hong Kong, Hong Kong, Hong Kong
- Hungary (4):
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Jávorszky Ödön Hospital, Vác
  - Csolnoky Ferenc Kórház, Veszprém
  - Zala County Hospital ICU, Zalaegerszeg
- Israel (11):
  - Haemek Medical Center, Afula
  - Soroka University Medical Centre, Beersheba
  - Wolfson Medical Center, Holon
  - Hadasit Medical Research Services and Development Ltd, Jerusalem
  - Galilee Medical Center, Nahariya
  - Nazareth EMMS Hospital, Nazareth
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - University Division of Infective and Tropical Diseases, University of Brescia, Italy, Brescia, Basilicate
  - Clinic of Infectious Diseases, Bologna, Emilia-Romagna
  - University Hospital Modena, Intensive Care Unit, Modena, Emilia-Romagna
  - National Institute for Infectious Diseases "L. Spallanzani", Rome, Lazio
  - Asst Di Cremona, Cremona, Lombardy
  - Ospedale San Raffaele - Milano, Milan, Lombardy
  - A.O.U. S. Giovanni di Dio e Ruggi d'Aragona, Salerno, Sardinia
- Mexico (6):
  - Hospital Civil de Guadalajara Dr Juan I Menchaca, Guadalajara
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Instituto Nacional de Ciencias; Medicas y Nutricion; Salvador Zubiran, Mexico City
  - CEPREP; Hospital Universitario, Monterrey
  - Hospital General de Tijuana, Tijuana
  - Centro de Especialidades Medicas Del Estado de Veracruz Dr Rafael Lucio, Xalapa
- Netherlands (8):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Gelre Ziekenhuizen Apeldoorn; Hospitals Pharmacy, Apeldoorn
  - LUMC, Leiden
  - UMC Radboud Nijmegen, Nijmegen
  - Erasmus Medical Centre; Department of Virology L-359, Rotterdam
  - Ikazia Hospital, Rotterdam
  - UMCU, Utrecht
  - Isala, Zwolle
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Tauranga Hospital, Tauranga
- Peru (13):
  - Hospital Regional del Cusco, Cusco
  - Hospital Nacional Adolfo Guevara Velasco, Cuzco
  - Hospital Guillermo Almenara Irigoyen Hospital Guillermo Almenara Irigoyen Hospital Guillermo Almen, La Victoria
  - Clinica Internacional Sede Lima, Lima
  - Hospital Nacional; Arzobispo Loayza, Lima
  - Hospital Nacional Hipolito; Unanue, Lima
  - Hospital Central Fuerza; Aerea del Peru, Lima
  - Hospital Maria Auxiliadora, Lima
  - Clínica San Gabriel, Lima
  - Clinica San Borja, Lima
  - Hospital de la Amistad Peru Corea II-2 Santa Rosa, Piura
  - Clinica Divino Nino Jesus; Orden de Malta, San Juán de Miraflores
  - Clinica Peruana Americana, Trujillo
- Poland (4):
  - Oddział Anestezjologii i Intensywnej Terapii Wojewódzki Specjalistyczny Szpital im dr Wł Biegańsk, Lodz
  - Wojewodzki Szpital Specjalistyczny, Lublin
  - Icu Spsk - 2, Szczecin
  - Oddział Anestezjologii i Intensywnej Terapii;Wojewódzki Szpital Zespolony im. L. Rydygiera, Torun
- Russia (4):
  - Municipal Clinical Hospital #8, Chelyabinsk
  - Municipal Healthcare Institution "City Hospital №2", Engel's
  - Medical Military Academy n.a S.M.Kirov, Saint Petersburg
  - Paciific state medical university, Vladivostok
- South Africa (3):
  - Milpark Hospital, Parktown West
  - Emmed Research, Pretoria
  - Clinical Projects Research, Worcester
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Gachon University Gil Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Yonsei University Health System/Severance Hospital, Seoul
  - Hallym university Kangnam Sacred Heart Hospital; Infectious devision, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (13):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Clinic, Barcelona, Cantabria
  - Hospital de Mataro, Mataro, Cantabria
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Bellvitge University Hospital, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Hosp. Clinico San Carlos, Madrid
  - Hospital Univ. de Getafe.Servicio de Neurologia, Madrid
  - Joan XXIII University Hospital, Tarragona
  - Servicio de Medicina Intensiva Hospital Universitario la Fe, Valencia
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Uppsala University Hospital, Department of Infectious Diseases, Gothenburg
  - Skånes Universitetssjukhus, Mamö
  - Norrland Universitetssjukhus, Umeå
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Cancer Center, Kaohsiung City
  - Far East Memorial Hospital, New Taipei City
  - Wanfang Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
- Ukraine (5):
  - Kyiv City Clinical Hospital #4, Kyiv
  - Kyiv City Clinical Hospital #9, Kyiv
  - Municipal Institution City Clinical Infectious Diseases Hospital, Odesa
  - Poltava Regional Clinical Infectious Hospital, Poltava
  - Municipal Institution Central City Hospital #1 City of Zhytomyr, Zhytomyr
- United Kingdom (9):
  - Queen Elizabeth Hospital, Birmingham
  - Heart of England NHS Trust, Birmingham
  - Queen Elizabeth University Hospital, Glasgow
  - Leeds General Infirmary, Anaesthetic Department, D Floor, Leeds
  - King College Hospital NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Southampton University Hospitals NHS Trust, Southampton
  - University Hospitals of North Midlands NHS Trust-Royal Stoke University Hospital, Stoke-on-Trent
  - Taunton and Somerset NHS Foundation Trust Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Lim JJ, Nilsson AC, Silverman M, Assy N, Kulkarni P, McBride JM, Deng R, Li C, Yang X, Nguyen A, Horn P, Maia M, Castro A, Peck MC, Galanter J, Chu T, Newton EM, Tavel JA. A Phase 2 Randomized, Double-Blind, Placebo-Controlled Trial of MHAA4549A, a Monoclonal Antibody, plus Oseltamivir in Patients Hospitalized with Severe Influenza A Virus Infection. Antimicrob Agents Chemother. 2020 Jun 23;64(7):e00352-20. doi: 10.1128/AAC.00352-20. Print 2020 Jun 23. PMID 32393496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled in the study were 168 participants. The participant flow is reported for the safety population (158 participants), which included all randomized participants who received study drug, with participants grouped according to the treatment actually received.
Groups:
- Placebo + Oseltamivir: Participants received a single IV dose of placebo matched to MHAA4549A on Day 1 and standard oseltamivir therapy for minimum of 5 days.
- MHAA4549A 3600 mg + Oseltamivir: Participants received a single low intravenous (IV) dose of MHAA4549A on Day 1 and standard oseltamivir therapy for minimum of 5 days.
- MHAA4549A 8400 mg + Oseltamivir: Participants received a single high IV dose of MHAA4549A on Day 1 and standard oseltamivir therapy for minimum of 5 days.
Period: Overall Study
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Started | 56 | 55 | 47
Completed | 47 | 42 | 38
Not Completed | 9 | 13 | 9
Not completed — Death | 4 | 6 | 4
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 3 | 1
Not completed — Reason Not Specified | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received study drug, with participants grouped according to the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir | Total
Number analyzed (Participants) | 56 | 55 | 47 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (17.5) | 56.5 (18.2) | 59.8 (17.9) | 60.7 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 22 | 71
  Male | 32 | 30 | 25 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 20 | 8 | 41
  Not Hispanic or Latino | 37 | 28 | 34 | 99
  Not Stated | 6 | 7 | 5 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 1 | 0 | 1 | 2
  Asian | 4 | 0 | 2 | 6
  Black or African American | 1 | 1 | 0 | 2
  White | 45 | 44 | 39 | 128
  Multiple | 0 | 1 | 0 | 1
  Unknown | 5 | 9 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: From randomization up to 60 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 56 | 55 | 47
percentage of participants | 80.4 | 67.3 | 74.5

2. Primary Outcome: Number of Participants With Anti-Therapeutic Antibodies (ATA) to MHAA4549A During and Following Administration of MHAA4549A
Description: Reported are the number of participants positive for ATAs at baseline, the number of participants with treatment-induced ATAs and the number of participants with treatment-enhanced ATAs.
Time Frame: From randomization up to 60 days
Population: Safety Population included all randomized participants who received study drug, with participants grouped according to the treatment actually received. Here, number analyzed are the participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 56 | 55 | 47
participants
  Positive for ATAs at baseline | 0 | 1 | 1
  Treatment-induced ATAs: number analyzed (Participants) | 47 | 43 | 37
  Treatment-induced ATAs | 0 | 0 | 0
  Treatment-enhanced ATAs: number analyzed (Participants) | 47 | 43 | 37
  Treatment-enhanced ATAs | 0 | 0 | 0

3. Primary Outcome: Time to Normalization of Respiratory Function
Description: The time to normalization of respiratory function was defined as the time to removal of the participant from oxygen (O2) supplementation in order to maintain a blood oxygen saturation level (SpO2) equal to or greater than 95% as measured by pulse oximetry.
Time Frame: From randomization up to 60 days
Population: Intent-to-treat infected (ITTi) population included all randomized participants who were confirmed to be influenza A infected, with participants grouped according to the treatment assigned at randomization.
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
days | 4.28 [3.06 to 6.60] | 2.78 [2.52 to 4.20] | 2.65 [1.58 to 4.52]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.6050, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.08, 80% CI 2-sided [0.83 to 1.40]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.2028, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.13, 80% CI 2-sided [0.85 to 1.51]

4. Secondary Outcome: Percentage of Participants by Clinical Status Using a Categorical Ordinal Outcome
Description: The clinical status of participants was defined by five mutually exclusive categories: 1. Death; 2. In the Intensive Care Unit (ICU); 3. Non-ICU hospitalization, requiring supplemental oxygen (O2); 4. Non-ICU hospitalization, not requiring supplemental oxygen (O2); 5. Not hospitalized.
Time Frame: Days 1-7, 14 and 30
Population: ITTi population included all randomized participants who were confirmed to be influenza A infected, with participants grouped according to the treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
percentage of participants
  Day 1: Death | 0.0 | 0.0 | 0.0
  Day 1: In ICU | 42.6 | 38.5 | 43.2
  Day 1: Non-ICU, requiring supplemental O2 | 57.4 | 61.5 | 52.3
  Day 1: Non-ICU, not requiring supplemental O2 | 0.0 | 0.0 | 4.5
  Day 1: Not hospitalized | 0.0 | 0.0 | 0.0
  Day 2: Death | 0.0 | 0.0 | 2.3
  Day 2: In ICU | 42.6 | 38.5 | 38.6
  Day 2: Non-ICU, requiring supplemental O2 | 40.7 | 51.9 | 31.8
  Day 2: Non-ICU, not requiring supplemental O2 | 11.1 | 7.7 | 20.5
  Day 2: Not hospitalized | 5.6 | 1.9 | 6.8
  Day 3: Death | 0.0 | 0.0 | 2.3
  Day 3: In ICU | 37.0 | 32.7 | 34.1
  Day 3: Non-ICU, requiring supplemental O2 | 31.5 | 42.3 | 27.3
  Day 3: Non-ICU, not requiring supplemental O2 | 20.4 | 19.2 | 25.0
  Day 3: Not hospitalized | 11.1 | 5.8 | 11.4
  Day 4: Death | 0.0 | 0.0 | 2.3
  Day 4: In ICU | 35.2 | 30.8 | 29.5
  Day 4: Non-ICU, requiring supplemental O2 | 25.9 | 21.2 | 18.2
  Day 4: Non-ICU, not requiring supplemental O2 | 22.2 | 36.5 | 29.5
  Day 4: Not hospitalized | 16.7 | 11.5 | 20.5
  Day 5: Death | 0.0 | 0.0 | 2.3
  Day 5: In ICU | 27.8 | 26.9 | 27.3
  Day 5: Non-ICU, requiring supplemental O2 | 25.9 | 19.2 | 18.2
  Day 5: Non-ICU, not requiring supplemental O2 | 24.1 | 34.6 | 27.3
  Day 5: Not hospitalized | 22.2 | 19.2 | 25.0
  Day 6: Death | 1.9 | 1.9 | 2.3
  Day 6: In ICU | 22.2 | 23.1 | 22.7
  Day 6: Non-ICU, requiring supplemental O2 | 22.2 | 15.4 | 15.9
  Day 6: Non-ICU, not requiring supplemental O2 | 27.8 | 34.6 | 25.0
  Day 6: Not hospitalized | 25.9 | 25.0 | 34.1
  Day 7: Death | 1.9 | 1.9 | 2.3
  Day 7: In ICU | 18.5 | 21.2 | 20.5
  Day 7: Non-ICU, requiring supplemental O2 | 24.1 | 13.5 | 15.9
  Day 7: Non-ICU, not requiring supplemental O2 | 14.8 | 28.8 | 25.0
  Day 7: Not hospitalized | 40.7 | 34.6 | 36.4
  Day 14: Death | 1.9 | 3.8 | 6.8
  Day 14: In ICU | 5.6 | 11.5 | 9.1
  Day 14: Non-ICU, requiring supplemental O2 | 7.4 | 3.8 | 6.8
  Day 14: Non-ICU, not requiring supplemental O2 | 14.8 | 3.8 | 4.5
  Day 14: Not hospitalized | 70.4 | 76.9 | 72.7
  Day 30: Death | 5.6 | 7.7 | 9.1
  Day 30: In ICU | 1.9 | 3.8 | 4.5
  Day 30: Non-ICU, requiring supplemental O2 | 5.6 | 1.9 | 4.5
  Day 30: Non-ICU, not requiring supplemental O2 | 1.9 | 3.8 | 0.0
  Day 30: Not hospitalized | 85.2 | 82.7 | 81.8

5. Secondary Outcome: Percentage of Participants With Clinical Failure
Description: Clinical failure after 24 hours post-infusion of study drug was defined as progression to increased O2 requirement defined by an increase in oxygen supplementation from low flow oxygen (i.e., 2-6 liters per minute [L/min]) to high flow oxygen (i.e., > 6 L/min) or from oxygen supplementation alone to any positive pressure ventilation (PPV) or extracorporeal membrane oxygenation (ECMO), progression to ICU, prolonged ventilation or O2 support defined by > 2 weeks, or death.
Time Frame: 24 hours after end of infusion (infusion duration = approximately 120 minutes) up to Day 60
Population: as for outcome 4
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
percentage of participants | 14.8 [8.82 to 22.95] | 25.0 [17.22 to 34.32] | 22.7 [14.63 to 32.84]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.1905, Cochran-Mantel-Haenszel; Difference in event rates = 10.19, 80% CI 2-sided [-0.15 to 20.52]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.3168, Cochran-Mantel-Haenszel; Difference in event rates = 7.91, 80% CI 2-sided [-2.64 to 18.47]

6. Secondary Outcome: Percentage of Participants With Clinical Resolution of Abnormal Vital Signs
Description: Description: Clinical resolution of abnormal vital signs was defined as meeting three out of five of the following criteria: 1. SpO2 ≥ 95% without supplemental O2; 2. Respiratory rate < 24 breaths per minute without supplemental O2; 3. Core temperature < 37.2 Celsius (C) immediately prior to receipt of any antipyretic drug, and at least 6-8 hours from the last dose of antipyretic or core temperature > 36 C in participants who are initially hypothermic; 4. Heart rate (HR) < 100 beats/minute; 5. Systolic blood pressure (SBP) >90 mmHg. Reported here is the percentage of participants who had clinical resolution of at least three out of five abnormal vital signs by the end of study.
Time Frame: From randomization up to 60 days
Population: as for outcome 4
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
percentage of participants | 81.3 [62.88 to 92.90] | 73.3 [53.60 to 87.82] | 66.7 [44.10 to 84.58]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.6043, Cochran-Mantel-Haenszel; Difference in event rates = -7.92, 80% CI 2-sided [-27.50 to 11.66]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.3865, Cochran-Mantel-Haenszel; Difference in event rates = -14.58, 80% CI 2-sided [-36.13 to 6.97]

7. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause
Time Frame: Days 14, 30 and 60
Population: as for outcome 4
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
percentage of participants
  Day 14 | 1.9 [0.19 to 7.01] | 3.8 [1.03 to 9.91] | 6.8 [2.53 to 14.56]
  Day 30 | 5.6 [2.06 to 11.95] | 7.7 [3.40 to 14.79] | 9.1 [4.02 to 17.35]
  Day 60 | 7.4 [3.27 to 14.26] | 9.6 [4.75 to 17.11] | 9.1 [4.02 to 17.35]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Day 14; Test type: Other; p = 0.5379, Cochran-Mantel-Haenszel; Difference in event rates = 1.99, 80% CI 2-sided [-5.57 to 9.56]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Day 14; Test type: Other; p = 0.2189, Cochran-Mantel-Haenszel; Difference in event rates = 4.97, 80% CI 2-sided [-3.12 to 13.05]
Statistical Analysis 3: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Day 30; Test type: Other; p = 0.6594, Cochran-Mantel-Haenszel; Difference in event rates = 2.14, 80% CI 2-sided [-6.04 to 10.31]
Statistical Analysis 4: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Day 30; Test type: Other; p = 0.5013, Cochran-Mantel-Haenszel; Difference in event rates = 3.54, 80% CI 2-sided [-5.24 to 12.31]
Statistical Analysis 5: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Day 60; Test type: Other; p = 0.6849, Cochran-Mantel-Haenszel; Difference in event rates = 2.21, 80% CI 2-sided [-6.28 to 10.69]
Statistical Analysis 6: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Day 60; Test type: Other; p = 0.7633, Cochran-Mantel-Haenszel; Difference in event rates = 1.68, 80% CI 2-sided [-7.38 to 10.74]

8. Secondary Outcome: Area Under Viral Load-Time Curve (AUEC ) of Influenza A Virus
Description: Influenza A viral load was measured by quantitative polymerase chain reaction (qPCR) in nasopharyngeal samples at multiple time points during the study. AUEC is the area under the viral load-time curve expressed as log10 (viral particles/milliliter x hour) = log10 (vp/mL x hour).
Time Frame: Immediately prior to MHAA4549A infusion and oseltamivir dosing on Day 1, immediately prior to oseltamivir dosing on Days 2 to 10, Days 14, 20, 25, 30, on day of discharge from hospital (up to Day 60), and at study completion (Day 60)
Population: ITTi population included all randomized participants who were confirmed to be influenza A infected, with participants grouped according to the treatment assigned at randomization. Here, number analyzed are the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: log10 (vp/mL x hour).
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 48 | 46 | 39
log10 (vp/mL x hour). | 25.72 (15.92) | 21.99 (16.57) | 25.03 (13.48)
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.2407, ANOVA; Mean Difference (Final Values) = -3.73, 80% CI 2-sided [-6.41 to -1.06]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.8339, ANOVA; Mean Difference (Final Values) = -0.70, 80% CI 2-sided [-3.49 to 2.10]

9. Secondary Outcome: Peak Influenza A Viral Load
Description: Influenza A viral load was measured by qPCR in nasopharyngeal samples at multiple time points during the study. Reported here is the peak Influenza A viral load expressed as log10 vp/mL.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: log10 vp/mL
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 48 | 46 | 39
log10 vp/mL | 5.70 (1.32) | 5.37 (1.39) | 5.28 (1.71)
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.2790, ANOVA; Mean Difference (Final Values) = -0.33, 80% CI 2-sided [-0.60 to -0.07]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.1909, ANOVA; Mean Difference (Final Values) = -0.42, 80% CI 2-sided [-0.70 to -0.15]

10. Secondary Outcome: Duration of Viral Shedding
Description: Influenza A viral load was measured by qPCR in nasopharyngeal samples at multiple time points during the study. Reported here is the duration of viral shedding.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
days | 4.00 [3.66 to 5.60] | 4.63 [3.63 to 4.97] | 4.60 [3.57 to 5.53]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.7413, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.01, 80% CI 2-sided [0.77 to 1.32]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.4763, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.32, 80% CI 2-sided [0.99 to 1.77]

11. Secondary Outcome: Duration of Hospitalization
Time Frame: From randomization up to 60 days
Population: as for outcome 4
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
days | 8.95 [5.90 to 10.29] | 7.65 [6.94 to 8.02] | 6.69 [6.00 to 8.86]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.8806, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.01, 80% CI 2-sided [0.78 to 1.32]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.5447, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.05, 80% CI 2-sided [0.80 to 1.38]

12. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Time Frame: From randomization up to 60 days
Population: as for outcome 8
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
days | 4.66 [3.91 to 7.10] | 6.60 [4.82 to 10.53] | 5.29 [3.25 to 6.58]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.4171, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.70, 80% CI 2-sided [0.47 to 1.03]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.8322, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.90, 80% CI 2-sided [0.61 to 1.34]

13. Secondary Outcome: Percentage of Participants Using Antibiotics for Respiratory Infections
Time Frame: From randomization up to 60 days
Population: as for outcome 4
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
percentage of participants | 13.0 [7.36 to 20.84] | 11.5 [6.17 to 19.37] | 11.4 [5.63 to 20.06]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.8240, Cochran-Mantel-Haenszel; Difference in event rates = -1.42, 80% CI 2-sided [-10.61 to 7.76]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.8111, Cochran-Mantel-Haenszel; Difference in event rates = -1.60, 80% CI 2-sided [-11.48 to 8.28]

14. Secondary Outcome: Percentage of Participants With Secondary Complications of Influenza
Description: The following were considered secondary complications of influenza: pneumonia, including hospital-acquired pneumonia (HAP) and ventilation-acquired pneumonia (VAP), exacerbations of chronic lung disease, myocarditis, acute respiratory distress syndrome (ARDS), otitis media, or other related complications.
Time Frame: From randomization up to 60 days
Population: as for outcome 4
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
percentage of participants | 13.0 [7.36 to 20.84] | 15.4 [9.17 to 23.79] | 13.6 [7.32 to 22.71]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.7219, Cochran-Mantel-Haenszel; Difference in event rates = 2.42, 80% CI 2-sided [-6.96 to 11.80]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.9225, Cochran-Mantel-Haenszel; Difference in event rates = 0.67, 80% CI 2-sided [-9.29 to 10.64]

15. Secondary Outcome: Percentage of Participants Readmitted to Hospital Due to Any Cause
Time Frame: Days 30 and 60
Population: as for outcome 4
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
percentage of participants | 1.9 [0.19 to 7.01] | 3.8 [1.03 to 9.91] | 0 [0.00 to 5.10]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.5379, Cochran-Mantel-Haenszel; Difference in event rates = 1.99, 80% CI 2-sided [-5.57 to 9.56]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.3667, Cochran-Mantel-Haenszel; Difference in event rates = -1.85, 80% CI 2-sided [-9.88 to 6.18]

16. Secondary Outcome: Duration of Ventilation
Time Frame: From randomization up to 60 days
Population: as for outcome 8
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 54 | 52 | 44
days | 4.11 [2.72 to 5.32] | 7.05 [1.92 to 13.12] | 5.89 [4.13 to 13.07]
Statistical Analysis 1: Comparison: Placebo + Oseltamivir vs MHAA4549A 3600 mg + Oseltamivir; Test type: Other; p = 0.7827, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.66, 80% CI 2-sided [0.41 to 1.07]
Statistical Analysis 2: Comparison: Placebo + Oseltamivir vs MHAA4549A 8400 mg + Oseltamivir; Test type: Other; p = 0.2522, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.58, 80% CI 2-sided [0.36 to 0.96]

17. Secondary Outcome: Area Under Serum Concentration-Time Curve From Time 0 to Infinity (AUC ) of MHAA4549A
Description: AUC0-inf is reported as day*microgram/milliliter (day*mcg/mL).
Time Frame: 30 minutes (min) before & 60 min after end of MHAA4549A infusion (infusion duration = 120 min) on Day 1; immediately prior to oseltamivir dose on Days 2, 3, 5, 7; on Days 14, 30; on day of discharge (up to Day 60); at study completion (Day 60)
Population: Pharmacokinetic (PK)-evaluable population included all participants, who received MHAA4549A and from whom evaluable PK samples were obtained.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 38 | 31
day*mcg/mL | 11400 (4530) | 26700 (9810)

18. Secondary Outcome: Maximum Serum Concentration (Cmax ) of MHAA4549A
Time Frame: 30 min before & 60 min after end of MHAA4549A infusion (infusion duration = 120 min) on Day 1; immediately prior to oseltamivir dose on Days 2, 3, 5, 7; on Days 14, 30; on day of discharge (up to Day 60); at study completion (Day 60)
Population: PK-evaluable population included all participants, who received MHAA4549A and from whom evaluable PK samples were obtained.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 38 | 31
mcg/mL | 916 (294) | 2220 (556)

19. Secondary Outcome: Elimination Half-Life (Terminal t1/2) of MHAA4549A
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: day
Arm/Group | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 38 | 31
day | 19.0 (4.91) | 17.8 (3.88)

20. Secondary Outcome: Observed Clearance (CL-obs) of MHAA4549A
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 38 | 31
mL/day | 288 (158) | 350 (130)

21. Secondary Outcome: Observed Steady State Volume of Distribution (Vss_obs) of MHAA4549A
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
Number analyzed (Participants) | 38 | 31
mL | 6410 (3170) | 7450 (2270)

ADVERSE EVENTS:
Time Frame: From randomization up to 60 days
Description: Safety Population included all randomized participants who received study drug, with participants grouped according to the treatment actually received.
Arm/Group | Placebo + Oseltamivir | MHAA4549A 3600 mg + Oseltamivir | MHAA4549A 8400 mg + Oseltamivir
All-Cause Mortality (participants affected / at risk) | 4/56 | 6/55 | 4/47
Serious Adverse Events (participants affected / at risk) | 8/56 | 11/55 | 12/47
Other Adverse Events (participants affected / at risk) | 28/56 | 26/55 | 18/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Oseltamivir (N=56) | MHAA4549A 3600 mg + Oseltamivir (N=55) | MHAA4549A 8400 mg + Oseltamivir (N=47)
Pneumonia (Infections and infestations) | 1 | 3 | 3
Septic shock (Infections and infestations) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 1
Ulcer (General disorders) | 0 | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Extubation (Surgical and medical procedures) | 0 | 0 | 1
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Oseltamivir (N=56) | MHAA4549A 3600 mg + Oseltamivir (N=55) | MHAA4549A 8400 mg + Oseltamivir (N=47)
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 1
Constipation (Gastrointestinal disorders) | 2 | 4 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypertension (Vascular disorders) | 7 | 1 | 4
Atrial fibrillation (Cardiac disorders) | 3 | 4 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 2
Pyrexia (General disorders) | 2 | 4 | 2
Agitation (Psychiatric disorders) | 4 | 3 | 1
Haematuria (Renal and urinary disorders) | 3 | 5 | 0
Headache (Nervous system disorders) | 2 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT02293863/Prot_SAP_000.pdf